CLINICAL TRIAL: NCT06343168
Title: Prevalence of Frailty and Associated Factors in Coronary Artery Bypass Patients
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Other Study IDs: frailty
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: prevalence of frailty — determine the prevalence of frailty

SUMMARY:
This study aimed to determine the prevalence of and factors affecting frailty in patients with coronary artery bypass graft.

The main question it aims to answer are:

What are the prevalence of and factors affecting frailty in patients with coronary artery bypass graft Type of study: descriptive cross-sectional study Participant population: coronary artery bypass grafting patients

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* planned CABG surgery
* volunteer to participate in the study

Exclusion Criteria:

* limb amputations
* stroke-related sequela
* hearing problems
* clinically unstable

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: coronary artery bypass grafting patients
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Prevalence of frailty | Preoperative
  Modified Fried Frailty Index

SECONDARY OUTCOMES:
Activities of Daily Living | Preoperative
  Barthel Activities of Daily Living Index
Nutritional Assessment | Preoperative
  Mini Nutritional Assessment Test-Short Form
Comorbidity | Preoperative
  Charlson Comorbidity Index
Cognitive Assessment | Preoperative
  Montreal Cognitive Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Usak University, Uşak, Center, Turkey (Türkiye)